CLINICAL TRIAL: NCT04820062
Title: Antibiotic Prescribing Behavior Among French Intensivist: Construction and Validation of a Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH031
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Antibiotic Reaction
Keywords: Antibiotic prescribing; questionnaire; Antibiotic resistance; behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Content Validity — For the validity of built, it is generally advisable to include a ratio of 100 participants for 30 questionnaire items. In order to have a suitable questionnaire, we will limit ourselves to 30 items which will be the size of our questionnaire. It was therefore planned to include 100 participants The selection of experts will be based on experience in this area, knowledge and availability. It will be a rescimant physician and an infectious disease doctor. Each expert will be invited in isolation to comment on the items in the questionnaire

SUMMARY:
Antibiotic resistance is a major threat in modern medicine. Overuse of antibiotics is an important driver of antibiotic resistance. However, some authors have shown that up to 50% of antibiotic treatments in critically ill patients are inappropriate, mostly because they are used in patients with non-bacterial infections.

In order to improve antibiotic use, several antibiotic stewardship programs have been implemented worldwide. However, only few of them have taken into account the determinants of prescribing behaviors. Yet, these determinants have been shown to play a role among general practitioners of hospital doctors. Nevertheless, none of these factors have been studied among intensivists.

The current project represent phase 1 of the study : construction and validation of a questionnaire.

DETAILED DESCRIPTION:
Antibiotic resistance is a major threat in modern medicine. Overuse of antibiotics is an important driver of antibiotic resistance. In critical care setting, antibiotic therapies are widely used due to the high number of patients presenting with sepsis. However, some authors have shown that up to 50% of antibiotic treatments in critically ill patients are inappropriate, mostly because they are used in patients with non-bacterial infections.

In order to improve antibiotic use, several antibiotic stewardship programs have been implemented worldwide. However, only few of them have taken into account the determinants of prescribing behaviors. Yet, these determinants have been shown to play a role among general practitioners of hospital doctors. Nevertheless, none of these factors have been studied among intensivists.

The study is designed to investigate social, cultural, contextual and personal factors influencing antibiotic prescribing among French intensivists. The design will consist of three phases:

* Phase 1: construction and validation of a questionnaire
* Phase 2: the questionnaire will be sent to all intensivist, including residents, in France
* Phase 3: qualitative study, based on semi-structured interviews.

The current project represent phase 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with predominant intensive care practice
* Resident, with a minimum of two-month experience in the intensive care unit

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians with predominant intensive care practice and Resident, with a minimum of two-month experience in the intensive care unit can be participe at this study.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Content validity | months 18
  Construction and validation of a questionnaire by 2 experts in reanimation and infectiology.
  This questionnaire will include these items: demographic datas, medical data concerning the use of antibiotics, social data exploring the collective and social components of antibiotic prescription, personal data in search of individual factors, attitude to antibiotic therapy.

SECONDARY OUTCOMES:
Face validity | months 18
  the questionnaire will be sent to all intensivist, including residents, in France

OTHER OUTCOMES:
Construct validity | months 18
  qualitative study, based on semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume THIERY, MD PHD, Principal Investigator — CHU ST ETIENNE FRANCE
Locations (1):
- Chu St Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No